CLINICAL TRIAL: NCT00922441
Title: A Randomized, Double-blind, Valsartan-Referenced, Parallel Grouped, Therapeutic Exploratory Clinical Study to Evaluate the Antihypertensive Efficacy of Fimasartan(BR-A-657•K) During 24hours by Dose in Patients With Mild to Moderate Essential Hypertension
Brief Title: A Therapeutic Exploratory Clinical Study to Evaluate the Antihypertensive Efficacy of Fimasartan (BR-A-657•K) During 24 Hours in Patients With Mild to Moderate Essential Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Collaborators: Seoul National University Hospital (Other); Kyungpook National University Hospital (Other); Catholic Medical Center (Other); Inje University (Other); Chonnam National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A657-BR-CT-203
Record Dates: First submitted 2009-06-16; First posted 2009-06-17 (Estimated); Results first posted 2018-02-13 (Actual); Last update posted 2018-03-15 (Actual); Status verified 2018-02

CONDITIONS: Essential Hypertension
Keywords: Fimasartan; Essential Hypertension; 24hour ABPM; Population PK
MeSH Terms: conditions — Essential Hypertension | interventions — fimasartan; Population Groups; Valsartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Fimasartan 1 (Experimental): Fimasartan 60 mg group
  Interventions: Drug: Fimasartan 60 mg group
- Fimasartan 2 (Experimental): Fimasartan 120 mg group
  Interventions: Drug: Fimasartan 120 mg group
- Valsartan (Active Comparator): Reference (Valsartan 80 mg) group
  Interventions: Drug: Reference (Valsartan 80 mg) group

INTERVENTIONS:
Drug: Fimasartan 60 mg group — Fimasartan 60 mg
  Other Names: BR-A-657.K
  Arms: Fimasartan 1
Drug: Fimasartan 120 mg group — Fimasartan 120 mg
  Other Names: BR-A-657.K
  Arms: Fimasartan 2
Drug: Reference (Valsartan 80 mg) group — Reference (Valsartan 80 mg)
  Other Names: Diovan
  Arms: Valsartan

SUMMARY:
The purpose of this study is to evaluate the antihypertensive efficacy and safety of Fimasartan (BR-A-657•K) during 24 hours by dose in patients with mild to moderate essential hypertension.

DETAILED DESCRIPTION:
Fimasartan(BR-A-657-K), a selective blocker of AT1 receptor subtype, showed the rapid and potent antihypertensive effect in many hypertensive models. Phase I study, Fimasartan(BR-A-657-K) 20mg ~ 480mg single dosing with healthy subjects, demonstrated that the Fimasartan(BR-A-657-K) was very safe and well tolerated. Another phase I study, Fimasartan(BR-A-657-K) 120mg and 360mg dosing for 7 days, also showed that Fimasartan(BR-A-657-K) was safe and tolerable though one temporal adverse event was observed in high dose.

A Randomized, Double-blind, Valsartan-referenced, Parallel Grouped, Therapeutic Exploratory Clinical Study to Evaluate the Antihypertensive Efficacy of Fimasartan(BR-A-657•K) during 24hoursby dose in Patients with Mild to Moderate Essential Hypertension.

Approximately 90 patients will be enrolled over 12 months in 5 centers nationwide.

After 2 weeks of placebo run-in period, all subjects will be randomized into one of the following 3 groups. Subjects will take test/control drug for 8 weeks of treatment period.

If subjects take any antihypertensive medications before screening, the subjects will have 1 week of wash-out period.

Group I : Fimasartan 60mg group. Group II : Fimasartan 120mg group Group III : Valsartan 80mg group

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate essential hypertension : sitting diastolic blood pressure measured at Placebo visit and Baseline are 90~109mmHg inclusive and the difference between sitting diastolic blood pressures measured at Placebo visit and Baseline(Day0) is under 7mmHg.
* Subjects who agree to participate in this sudy and give written informed consent
* Subjects considered to understand the study, be cooperative, and able to be followed-up until the end of the study

Exclusion Criteria:

* The sitting DBP is less than 89mmHg or more than 110mmHg or severe hypertensive patient with sitting systolic blood pressure over 200mmHg Patients with secondary hypertension
* Patients with severe renal(Creatinine more 1.5mg/dl), gastrointestinal, hematological or hepatic(AST, ALT more 2 twice more than upper limit of normal)disease etc. which might affect absorption, disposition, metabolism or excretion of the drug
* Patients with postural hypotension
* Patients with sever insulin dependent diabetes mellitus or uncontrolled diabetes mellitus(HbA1c>9%, regimen change of oral hypoglycemic agents within 12weeks, treated insulin before screening)
* Patients with a history of myocardial infarction, severe coronary artery disease or clinically significant heart failure or valvular defect in last 6 months
* Patients with consumptive disease, autoimmune disease, connective tissue disease
* Patients with a history of type B or C hepatitis
* Patients with HIV or hepatitis
* Patients with clinically significant laboratory abnormality
* Patients receiving any drugs known to affect blood pressure or medical treatments that can influence the blood pressure
* Patients with allergy or contraindication to any angiotensin II receptor antagonists
* Female of childbearing potential who does not undergo hysterectomy or is not post-menopausal
* Patients judged to have a history of alcohol or drug abuse by the investigator
* Patients participated other clinical trial 12 weeks before Screening Patients judged to be inappropriate for this study by the investigator with other reasons

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2008-12; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Byung-He Oh, Professor, Study Chair — Seoul National University Hospital; Dong-Soo Kim, Professor, Principal Investigator — Inje University; Sung Chul Chae, Professor, Principal Investigator — Kyungpook National University Hospital; Gi-Sik Kim, professor, Principal Investigator — Daegu Catholic University Medical Center; Myung-Ho Jung, Professor, Principal Investigator — Connam National University Hospital

REFERENCES:
- [Derived] Lee H, Kim KS, Chae SC, Jeong MH, Kim DS, Oh BH. Ambulatory blood pressure response to once-daily fimasartan: an 8-week, multicenter, randomized, double-blind, active-comparator, parallel-group study in Korean patients with mild to moderate essential hypertension. Clin Ther. 2013 Sep;35(9):1337-49. doi: 10.1016/j.clinthera.2013.06.021. Epub 2013 Aug 7. PMID 23932463

RESULTS

PARTICIPANT FLOW:
Groups:
- Fimasartan 1: Fimasartan 60 mg group
  Fimasartan 60 mg daily, po
- Fimasartan 2: Fimasartan 120 mg group
  Fimasartan 120 mg daily, po
- Valsartan: Control: Reference (Valsartan 80 mg) group
  Valsartan 80 mg daily, po
Period: Overall Study
Arm/Group | Fimasartan 1 | Fimasartan 2 | Valsartan: Control
Started | 30 | 30 | 32
Completed | 30 | 30 | 29
Not Completed | 0 | 0 | 3
Not completed — Protocol Violation | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fimasartan 1 | Fimasartan 2 | Valsartan: Control | Total
Number analyzed (Participants) | 30 | 30 | 32 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.07 (8.36) | 54.07 (8.79) | 56.00 (7.15) | 54.09 (8.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 14 | 13 | 36
  Male | 21 | 16 | 19 | 56

OUTCOME MEASURES:

1. Primary Outcome: Mean Change of Diastolic Blood Pressure
Description: 24hr Mean change of DBP on Week 8, from Baseline
Time Frame: baseline and 8 Weeks
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Fimasartan 1-ITT: Fimasartan 60 mg group
  Fimasartan 60 mg daily, po
- Fimasartan 2-ITT: Fimasartan 120 mg group
  Fimasartan 120 mg daily, po
- Valsartan: Control-ITT: Reference (Valsartan 80 mg) group
  Valsartan 80 mg daily, po
Arm/Group | Fimasartan 1-ITT | Fimasartan 2-ITT | Valsartan: Control-ITT
Number analyzed (Participants) | 30 | 30 | 29
mmHg | -10.15 (5.94) | -7.19 (9.51) | -6.70 (6.61)
Statistical Analysis 1: Comparison: Fimasartan 1-ITT vs Fimasartan 2-ITT vs Valsartan: Control-ITT; Test type: Other — Efficacy, Safety; p < 0.05, ANOVA; comparison between the groups

ADVERSE EVENTS:
Arm/Group | Fimasartan 1 | Fimasartan 2 | Valsartan: Control
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/32
Other Adverse Events (participants affected / at risk) | 4/30 | 5/30 | 2/32
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fimasartan 1 (N=30) | Fimasartan 2 (N=30) | Valsartan: Control (N=32)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
ALT Increased (Investigations) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No